CLINICAL TRIAL: NCT05193500
Title: Study 3 Learning Verbs and Pronouns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: Emerson College (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 280523
Record Dates: First submitted 2022-01-03; First posted 2022-01-18 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verbs (Experimental): Children hear a novel verb in an experimental context that is personally relevant to them (e.g., addressed, of interest) or neutral.
  Interventions: Behavioral: Verbs
- Pronouns (Experimental): Children hear a pronoun in an experimental context that is personally relevant to them (e.g., addressed, of interest) or neutral.
  Interventions: Behavioral: Pronouns

INTERVENTIONS:
Behavioral: Verbs — New verbs are introduced that are personally relevant to the child or neutral.
  Arms: Verbs
Behavioral: Pronouns — Pronouns are used that directly refer to the child or are neutral.
  Arms: Pronouns

SUMMARY:
The goal of this research is to explore abilities to learn word meanings from overheard speech in children with ASD (and, as a control, typically developing children).

Specific Aim 3 (Experiment 3): Determine whether children with ASD can learn verbs and pronouns by overhearing. Most prior work on learning from overheard speech has focused on learning nouns that label objects. This experiment extends this work to study other kinds of words.

ELIGIBILITY:
Inclusion Criteria:

* children with or without a diagnosis of ASD between 24 to 71 months of age

Exclusion Criteria:

* native language is not English
* born premature (< 36 weeks)
* has uncorrected hearing or vision impairments
* has developmental disorders or medical conditions other than ASD that affect language or cognition (excepting psychiatric conditions often comorbid with ASD such as ADHD)
* has a history of photosensitive epileptic seizures

Ages: 24 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 179 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-01-05 (Actual); Study Completion 2025-01-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Emerson College, Boston, Massachusetts
  - New York University, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- ASD - Verbs: Children with ASD hear a novel verb in an experimental context that is personally relevant to them (e.g., addressed, of interest) or neutral.
- ASD - Pronouns: Children with ASD hear a pronoun in an experimental context that is personally relevant to them (e.g., addressed, of interest) or neutral.
- TD - Verbs: Children with TD hear a novel verb in an experimental context that is personally relevant to them (e.g., addressed, of interest) or neutral.
- TD - Pronouns: Children with TD hear a pronoun in an experimental context that is personally relevant to them (e.g., addressed, of interest) or neutral.
Period: Overall Study
Arm/Group | ASD - Verbs | ASD - Pronouns | TD - Verbs | TD - Pronouns
Started | 75 | 13 | 67 | 23
Completed | 68 | 9 | 64 | 18
Not Completed | 7 | 4 | 3 | 5
Not completed — Withdrawal by Subject | 7 | 4 | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- ASD - Verbs; TD - Verbs: Children hear a novel verb in an experimental context that is personally relevant to them (e.g., addressed, of interest) or neutral.
- ASD - Pronouns; TD - Pronouns: Children hear a pronoun in an experimental context that is personally relevant to them (e.g., addressed, of interest) or neutral.
- Total: Total of all reporting groups
Arm/Group | ASD - Verbs | TD - Verbs | ASD - Pronouns | TD - Pronouns | Total
Number analyzed (Participants) | 75 | 67 | 13 | 23 | 178
Age, Continuous [Mean (Standard Deviation); unit: months] | 56.7 (11.0) | 37.5 (12.2) | 61.3 (11.0) | 45.5 (9.4) | 49.3 (14.3)
Sex/Gender, Customized [Number; unit: participants]
  Number of Enrolled Males | 57 | 48 | 6 | 22 | 133
  Number of Enrolled Females | 18 | 19 | 7 | 1 | 45
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 3 | 3 | 3 | 10
  Black | 10 | 0 | 1 | 0 | 11
  More than one race | 13 | 12 | 4 | 8 | 37
  Hispanic | 4 | 0 | 0 | 0 | 4
  Unknown | 4 | 2 | 1 | 4 | 11
  White | 43 | 50 | 4 | 8 | 105
Region of Enrollment [Number; unit: participants]
  United States | 75 | 67 | 13 | 23 | 178

OUTCOME MEASURES:

1. Primary Outcome: Object Preference for Verbs
Description: Proportion of Time During Which Children's Eye Gaze is Directed Toward the Target Object in the Window from 1.0-2.5 Seconds after the Test Question
Time Frame: During test phase of the experimental session (within 3 seconds after the learning phase); 1.0-2.5 seconds after the test question
Population: Participants were excluded from this outcome variable if their data was not able to be reliably coded (e.g., children were not looking at the screen).
Measure: Mean (Standard Deviation); unit: proportion of time
Arm/Group | ASD - Verbs | TD - Verbs
Number analyzed (Participants) | 60 | 60
proportion of time | 0.57 (0.29) | 0.56 (0.22)
Statistical Analysis 1: Comparison: ASD - Verbs; Test type: Other; p = 0.085, t-test, 2 sided — a priori threshold for statistical significance is 0.05; one-sample t-test, compared to 0.5 (chance)
Statistical Analysis 2: Comparison: TD - Verbs; Test type: Other; p = 0.049, t-test, 2 sided — a priori threshold for statistical significance is 0.05

2. Primary Outcome: Object Selection for Pronouns
Description: Proportion of trials on which children select the correct object that matches the pronoun
Time Frame: During test phase of the experimental session (within approx. 5 seconds of being asked the test question)
Population: Participants were excluded from this outcome variable if their data was not able to be reliably coded (e.g., children selected multiple objects at the same time).
Measure: Mean (Standard Deviation); unit: Proportion of correct object selections
Units Other Than Participants: trials
Arm/Group | ASD - Pronouns | TD - Pronouns
Number analyzed (Participants) | 7 | 17
Number analyzed (trials) | 53 | 131
Proportion of correct object selections | 0.67 (0.13) | 0.84 (0.15)
Statistical Analysis 1: Comparison: ASD - Pronouns vs TD - Pronouns; Test type: Other; p = 0.015, t-test, 2 sided — a priori threshold for statistical significance = 0.05

ADVERSE EVENTS:
Time Frame: 2 years, 5 months
Description: Our experimental paradigm involves presenting children with everyday child-friendly actions during a 10-minute interaction. There is no risk of Serious Adverse Events or All-Cause Mortality during the session.
Arm/Group | ASD - Verbs | TD - Verbs | ASD - Pronouns | TD - Pronouns
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/67 | 0/13 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/67 | 0/13 | 0/23
Other Adverse Events (participants affected / at risk) | 0/75 | 0/67 | 0/13 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT05193500/Prot_SAP_001.pdf
  • Informed Consent Form (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/00/NCT05193500/ICF_000.pdf